CLINICAL TRIAL: NCT05942001
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of HRS-5041 in Subjects With Metastatic Castration-resistant Prostate Cancer
Brief Title: Study of HRS-5041 in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5041-101
Record Dates: First submitted 2023-07-05; First posted 2023-07-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Advanced Prostate Cancer

STUDY DESIGN:
Intervention Model Description: HRS-5041 single arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-5041 (Experimental)
  Interventions: Drug: HRS-5041

INTERVENTIONS:
Drug: HRS-5041 — HRS-5041 was given oral administration, qd, at a 28-day cycle. Patients may continue to use HRS-5041 until disease progression or unacceptable toxicity occurs.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and preliminary efficacy of HRS-5041 in men with progressive metastatic castration resistant prostate cancer. The objective of this study was to determine the dose-limiting toxicity, maximum tolerance and recommended dose of HRS-5041 in phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Age 18-80 years old, gender unlimited.
3. The physical status score of the Eastern Tumor Cooperative Group (ECOG) was 0 ~ 1.
4. Predicted survival ≥12 weeks.
5. Histological or cytological confirmed adenocarcinoma of the prostate.
6. Patients progressed on taxane chemotherapy and at least one prior secondary hormonal therapy.

Exclusion Criteria:

1. Prior treatment with an androgen receptor (AR) degrader.
2. Plan to receive any other antitumor therapy during this trial.
3. Receiving other investigational drugs or treatments that are not on the market within 4 weeks prior to the initial administration of the study.
4. Patients with known brain metastases.
5. Any significant medical condition, such as uncontrolled infection, laboratory abnormality, or psychiatric illness.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days
Maximum tolerated dose (MTD) | Up to 28 days
Recommended Phase 2 Dose (RP2D) of HRS-5041 | Up to 28 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) evaluated using the NCI CTCAE v5.0 criteria | From the time of consent at screening until 30 days after the subject discontinues study treatment, up to 2 years
Pharmacokinetics - Area under the plasma concentration time curve (AUC) | 12 weeks
Pharmacokinetics - Maximum plasma concentration (Cmax) | 12 weeks
Pharmacokinetics - Time to Cmax (Tmax) | 12 weeks
Prostate Specific Antigen (PSA) decline of ≥ 50% from baseline (PSA50) | 24 months
PSA Progression Free Survival (PFS) | 24 months
Objective soft tissue response defined by complete response (CR) or partial response (PR) per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) | 24 months
Radiographic progression free survival (rPFS) | 24 months
Overall survival (OS) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided